CLINICAL TRIAL: NCT05861362
Title: Feasibility and Metabolic Effects of a 5:2 Fasting Intervention in Women With Breast Cancer During Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MVZ Leopoldina GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-01
Record Dates: First submitted 2023-05-02; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAST (Experimental): 5:2 intermittent fasting group
  Interventions: Radiation: Curative radiotherapy; Behavioral: 5:2 intermittent fasting

INTERVENTIONS:
Radiation: Curative radiotherapy — Curative radiotherapy as indicated by the patient's disease and prescribed by the treating radiation oncologist
Behavioral: 5:2 intermittent fasting — Two nonconsecutive days of fasting per week that could be chosen freely according to the patient's weekly schedule.

SUMMARY:
The intervention consists of the adoption of a 5:2 intermittent fasting diet during radiotherapy of breast cancer patients. The aim of the study was to assess the feasibility of this intervention and its impact on body composition and selected metabolic blood parameters.

DETAILED DESCRIPTION:
The 5:2 intermittent fasting (FAST) intervention consisted of two nonconsecutive days of fasting per week that could be chosen freely according to the patient's weekly schedule. The minimum amount of time to count as a fasting day was 24 hours, but patients were advised to aim for a complete fasting day including the nights before and after that day. On a fasting day, only water and unsweetened tea or coffee was allowed. However, given that fat is the macronutrient interfering the least with the metabolic adaptions to fasting, while carbohydrates disturb the most [26], patients were allowed to consume small amounts of bone broth/meat broth, coconut oil, butter/ghee or heavy cream as an "emergency plan", i.e., in case that they felt they needed some energy-containing foods to complete an initiated fasting day.

The primary study outcome was the feasibility of the FAST intervention and its effects on longitudinal body composition changes from baseline until the final week of radiotherapy (body mass, fat mass, fat-free mass, muscle mass, extracellular and total body water). Secondary endpoints were absolute changes in metabolic parameters, hormones, and overall quality of life scores in the FAST group. As a surrogate marker for insulin resistance, the triglyceride-glucose index (TyG) was calculated according to TyG=ln⁡(fasting triglycerides [mg/dl]×fasting glucose [mg/dl]/ 2).

ELIGIBILITY:
Inclusion Criteria:

* Non-metastasized breast cancer
* Indication for curative radiotherapy

Exclusion Criteria:

* metallic body parts that would interfere with electric bioimpedance (BIA) measurements
* difficulties with understanding the aims of the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Dropout rate in the FAST intervention group | Through study completion, an average of 5 weeks
  Used to measure feasibility. The intervention is rated as feasible if dropout rate is <30%
Longitudinal changes in body mass | Through study completion, an average of 5 weeks
  Body mass (in kg) is measured by a bioimpedance device with an integrated scale (seca mBCA, seca Deutschland, Hamburg, Germany).
Longitudinal changes in fat-free mass | Through study completion, an average of 5 weeks
  Fat-free mass (in kg) is estimated by a bioimpedance device with an integrated scale (seca mBCA, seca Deutschland, Hamburg, Germany).
Longitudinal changes in skeletal muscle mass | Through study completion, an average of 5 weeks
  Skeletal muscle mass (in kg) is estimated by a bioimpedance device with an integrated scale (seca mBCA, seca Deutschland, Hamburg, Germany).
Longitudinal changes in total body water | Through study completion, an average of 5 weeks
  Total body water content (in L) is estimated by a bioimpedance device with an integrated scale (seca mBCA, seca Deutschland, Hamburg, Germany).
Longitudinal changes in extracellular water | Through study completion, an average of 5 weeks
  Extracellular water (in L) is estimated by a bioimpedance device with an integrated scale (seca mBCA, seca Deutschland, Hamburg, Germany).

SECONDARY OUTCOMES:
Change between baseline and final (average 5 weeks) TyG index | Through study completion, an average of 5 weeks
  As a surrogate marker for insulin resistance, the triglyceride-glucose index (TyG) is calculated according to TyG=ln⁡(fasting triglycerides [mg/dl]×fasting glucose [mg/dl]/ 2)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer J Klement, Ph.D., Principal Investigator — Department of Radiation Oncology, Leopoldina Hospital Schweinfurt
Locations (2):
- Germany (2):
  - Department of Radiotherapy and Radiation Oncology, Schweinfurt, Bavaria
  - Leopoldina Hospital Schweinfurt, Department of Radiotherapy and Radiation Oncology, Schweinfurt, Bavaria

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request